CLINICAL TRIAL: NCT03690726
Title: The Effects of Systematic, Repetitive Transcranial Magnetic Stimulation in Rehabilitation After Incomplete Spinal Cord Injury: Neuromuscular Adaptations and Recovery of Lower Limb Muscle Strength
Brief Title: The Effects of rTMS in Rehabilitation Following Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spinal Cord Injury Centre of Western Denmark (Other)
Collaborators: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Helge Kasch, Medical Research Director, Associate Professor, Clinical Neurology, MD, PhD, Spinal Cord Injury Centre of Western Denmark
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VCR-rTMS
Record Dates: First submitted 2018-09-20; First posted 2018-10-01 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Spinal Cord Injury; Rehabilitation; Transcranial Magnetic Stimulation; Neurorehabilitation
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Randomized Placebo Controlled Clinical Intervention Study
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active rTMS (Experimental): SCI patients fulfilling criteria for participation giving informed written and verbal consent, who are enrolled and randomised to active treatment arm receive consecutive treatment sessions with rTMS directed at cranium and cortex regions as described in protocol.
  Interventions: Device: repetitive transcranial magnetic stimulation
- Sham rTMS (Sham Comparator): SCI patients fulfilling criteria for participation giving informed written and verbal consent, who are enrolled and randomised to sham/control arm receive consecutive treatment sessions with coil from rTMS that fires at other spot (pillow/mattress) as described in protocol.
  Interventions: Other: Sham stimulation

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation — Repetitive transcranial magnetic stimulation of the leg motor cortex, in combination with resistance training
  Arms: Active rTMS
Other: Sham stimulation — Imitated magnetic stimulation: An active coil will be activated under the subject's head, firing down into the mattress, while an inactive coil will be held over the scalp
  Arms: Sham rTMS

SUMMARY:
The project will investigate whether repetitive transcranial magnetic stimulation (rTMS) can be used to potentiate/prime spinal cord injured patients' nervous systems for more intense rehabilitation exercise of longer duration - thus leading to greater recovery of motion function. The technique, in which a magnetic coil is positioned above the scalp and forms a magnetic field that activates the desired center of the brain (eg motor cortex), is used in clinical practice for the treatment of a number of disorders. However, although a combination of rTMS and gait training in SCI patients previously has proven beneficial, it is unknown whether additional functional gains can be achieved by combining rTMS and supervised, high-intensity resistance training.

In this project, 30 newly-admitted patients will be recruited and randomized to receive either active rTMS and strength training (n = 15) or sham (imitated) rTMS + strength training, in parallel with standard care. The investigators hypothesize that the active rTMS group will have superior gains in locomotor function and muscle mass, compared to the sham group.

ELIGIBILITY:
Inclusion Criteria:

* sub-acute (<6 months) incomplete spinal cord injury
* admitted at the SCIWDK for primary rehabilitation

Exclusion Criteria:

* Medical history of multiple central nervous system lesions,
* severe structural,
* inflammatory or degenerative cerebral disorders,
* epilepsy,
* other neurological diseases,
* lower limb peripheral injury,
* or orthopedic injuries that may limit maximal effort contractions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
6 minutes walking test | Measures the change from baseline and after 8 weeks of intervention
  Test of ambulatory endurance. It measures the maximal distance covered within 6 minutes.
Lower limb maximal muscle strength | Measures the change from baseline and after 8 weeks of intervention
  Measures the maximal voluntary contraction torque of the knee flexors and knee extensors.
Timed up and go test | Measures the change from baseline and after 8 weeks of intervention
  Measures the time (in seconds) it takes a person to get up from an ordinary chair with back and armrest, walk 3 meters, turn back to the chair and sit back.
Rate of force development | Measures the change from baseline and after 8 weeks of intervention
  Measures the explosive muscle force of the knee flexors and knee extensors.
10 meter walking test | Measures the change from baseline and after 8 weeks of intervention
  Measures the time (in seconds) it takes to cover 10 meters during level-ground walking.

SECONDARY OUTCOMES:
Quantitative Sensory Testing | Measures the change from baseline and after 8 weeks of intervention
  Measures the sensitivity to heat and cold stimuli on the skin.
H-reflex test | Measures the change from baseline and after 8 weeks of intervention
  Measures spasticity from the ratio of the amplitude between the M-wave and H-wave. These are evoked during a short electrical stimulation impulse delivered to the nerves innervating the soleus muscle.
Modified Ashworth Scale | Measures the change from baseline and after 8 weeks of intervention
  A manual test that measures spasticity from 0 to 4, where 0 is no spasticity and 4 is widespread spasticity.
The International Standards for Neurological Classification of Spinal Cord Injury | Measures the change from baseline and after 8 weeks of intervention
  An examination that is used to score the motor and sensory impairment and severity of a spinal cord injury.
Walking Index for Spinal Cord Injury test | Measures the change from baseline and after 8 weeks of intervention
  A test that assesses the amount of physical assistance needed, as well as devices required, for walking following paralysis that results from Spinal Cord Injury.
Pressure algometry | Measures the change from baseline and after 8 weeks of intervention
  A test for the pressure sensitivity of the pain nerve fibers in and superficial to the masseter and soleus muscles.
Self-reported pain | Measures the change from baseline and after 8 weeks of intervention
  Examines self-reported pain through a 100mm Visual-Analogue Scale, scored 0-100, where 0 is "no pain" and 100 is "the greatest pain imaginable".

CONTACTS AND LOCATIONS:
Overall Officials: Helge Kasch, MD, PhD, Principal Investigator — Spinal Cord Injury Centre of Western Denmark
Locations (1):
- Spinal Cord Injury Centre of Western Denmark, Viborg, Denmark

IPD SHARING:
Plan to Share IPD: No